CLINICAL TRIAL: NCT05849818
Title: Virtual Reality Technology For Cognitive Functions Of Children With Down Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ayman Kamal Elboraey, Professor of Pediatric physical therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ayman Kamal
Record Dates: First submitted 2023-04-14; First posted 2023-05-09 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-04

CONDITIONS: Down Syndrome
Keywords: Down syndrome DS; Virtual Reality VR
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Intervention Model Description: A prospective Randomized controlled trial of pre-post study design with a two months follow up evaluation will be used
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Effect of fully immersive VR + school regular activities on cognitive functions of Down children (Experimental): Children in this group will practice the same activities as control group in addition to virtual reality session using fully-immersive VRapeutic software gaming technology (Viblio module)for 20 min/3sessions/week for 8 weeks.
  Interventions: Device: full-immersive VRapeutic software gaming technology
- Effect of school regular activities on cognitive functions of down children (No Intervention): Children in this group will practice their regular activities of school and daily living (receive no treatment).

INTERVENTIONS:
Device: full-immersive VRapeutic software gaming technology — * Children of the study group will receive VR training sessions 3 times per week for 8 successive weeks.
  * Viblio VRapeutic fully immersive game will be used.
  * Manual instructions of the game will be followed and features of the game will be customized.
  * The child instructed to put back a pile of books on the floor into their shelves.
  * Level II of the game we will use audio visual distractors , repeated parrot sound and the child is required to order the books by colors
  * Level III distracting tasks during book ordering
  * The complexity of the game depend on task duration, number of books and the nature of distractors
  Other Names: VRapeutic software gaming technology
  Arms: Effect of fully immersive VR + school regular activities on cognitive functions of Down children

SUMMARY:
The purpose of the study is to identify the effect of fully-immersive virtual reality technology on cognitive functions of children with Down syndrome

DETAILED DESCRIPTION:
Intellectual disability is recognized as one of the most prominent features of DS which is the most common genetic cause of intellectual disability. Cognitive functioning often changes across the lifespan and is moderated by several comorbid factors such as sensory impairments, seizures, autism, sleep disruption, and other medical and psychiatric conditions (Grieco et al., 2015).

There is encouraging evidence supporting the use of non-immersive virtual environments to provide useful learning, rehabilitation, and leisure experiences for people with intellectual disabilities. Therefore, immersive VR applications may also be an effective way to improve motivation and engagement for children with DS in learning settings (Michalski et al., 2022). Therefore, this study aims to investigate the effect of full-immersive VRapeutic software gaming technology on cognitive functions of children with Down syndrome

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Down Syndrome Age from 6-10 years Both Genders will be included IQ Ranges from 50-69(mild intellectual disability) they will be able to understand the instructions able to walk independently

Exclusion Criteria:

* Significant Visual or Hearing problems Significant mental or psychological problems that interfere with understanding instructions musculoskeletal problems or fixed deformities in upper or lower limbs Current hospitalization for urgent Medical reasons

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Rate of change of cognitive function by using the rehacom device | up to two months
  Assessing the change of the cognitive function By using the Rehacom Device within two months

CONTACTS AND LOCATIONS:
Overall Officials: Amira Eltohamy, professor, Principal Investigator — Cairo University
Locations (1):
- Cairo University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No